CLINICAL TRIAL: NCT04865835
Title: A Randomized, Single-blind, Two-period Crossover to Investigate the Effect of SEP-363856 on the Pharmacokinetics of Metformin in Subjects With Schizophrenia.
Brief Title: A Clinical Trial Study to Determine the Effect of an Investigational Drug (SEP-363856) Has on the Way That the Drug Metformin Travels Through the Body in People With Schizophrenia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SEP361-110
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856; Metformin

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, two-period crossover study in adults with schizophrenia
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo and metformin (Placebo Comparator): single dose of placebo + single dose of metformin-HCl 850 mg (approximately 663 mg metformin) (placebo will be dosed 1 hour prior to metformin administration)
  Interventions: Drug: placebo; Drug: metformin
- SEP-363856 and metformin (Experimental): single dose of SEP 363856 100 mg + single dose of metformin-HCl 850 mg (SEP 363856 will be dosed 1 hour prior to metformin administration)
  Interventions: Drug: SEP-363856; Drug: metformin

INTERVENTIONS:
Drug: placebo — single dose of placebo
  Arms: placebo and metformin
Drug: SEP-363856 — single dose of SEP 363856 100 mg
  Arms: SEP-363856 and metformin
Drug: metformin — metformin-HCl 850 mg

SUMMARY:
A clinical trial study to determine the effect of an investigational drug (SEP-363856) has on the way that the drug Metformin travels through the body in people with schizophrenia. This clinical trial will have approximately 24 subjects both male and female 18 year of age and older. This study will be conducted in approximately 2 study sites in the United States.

DETAILED DESCRIPTION:
This is a randomized, single-blind, two-period crossover study in which each subject will receive both treatments and therefore act as their own control to minimize confounding covariates within the study population. Randomizing subjects to treatment sequence will assist with reducing the potential order effects that might confound the findings if all the subjects received the same treatment sequence. The single-blind method is used to keep subjects blind to treatment assignment throughout the study period, in order to avoid possible influence of the psychological factors of subjects on study assessments. This clinical study will evaluate whether SEP 363856 influences the PK of a concomitantly administered OCT2 substrate, metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 65 years of age, inclusive, at the time of informed consent.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM 5) criteria for a primary diagnosis of schizophrenia as established by clinical interview (using the DSM 5 as a reference and confirmed using the Structured Clinical Interview for DSM 5, Clinical Trials Version [SCID CT]).
* Subject must have a Clinical Global Impressions - Severity Scale (CGI S) score ≤ 4 (normal to moderately ill) at Screening.
* Subject must have a Positive and Negative Syndrome Scale (PANSS) total score ≤ 80 at Screening.
* Subject must have a score of ≤ 4 on the following PANSS items at Screening:

P7 (hostility) G8 (uncooperativeness).

* Subject must have normal to mild symptoms on all individual items of the Simpson-Angus Scale (SAS) (< 2), Abnormal Involuntary Movement Scale (AIMS) (< 3) and Barnes Akathisia Rating Scale (BARS) (< 3) at Screening.
* Subject has been taking an antipsychotic for at least six weeks prior to Screening and has had no change in antipsychotic medication(s) (minor dose adjustments for tolerability purposes may be permitted after Medical Monitor and Sponsor review) for at least six weeks prior to Screening.

Exclusion Criteria:

* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study, including any clinically significant hematological (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urological, cardiovascular, hepatic, neurologic or allergic disease (except for untreated seasonal allergies that are asymptomatic at the time of dosing).

  * Subject has a disorder or history of a condition, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection) that may interfere with drug absorption, distribution, metabolism, excretion, gastrointestinal motility, or pH, or a history of clinically significant abnormality of the hepatic or renal system, or a history of malabsorption (uncomplicated cholecystectomy, appendectomy, and hernia repair will be acceptable).
  * Subject has a DSM 5 diagnosis or presence of symptoms consistent with a DSM 5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms are not the primary focus of treatment.
  * Subject answers "yes" to "Suicidal Ideation" Items 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the Columbia-Suicide Severity Rating Scale (C SSRS) at Screening (ie, in the past 1 month) or at any subsequent C SSRS assessment prior to dosing (ie since last visit).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | 72 hours
  area under the plasma concentration-time curve from time zero to infinity (AUC0 ∞) or area under the plasma concentration-time curve from time zero to a defined time (AUC0-t), if appropriate
• maximum observed plasma concentration | 72 hours
  maximum observed plasma concentration (Cmax).

SECONDARY OUTCOMES:
area under the plasma concentration-time curve | 72 hours
  area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (AUC0-last)
time of the maximum observed plasma concentration | 72 hours
  time of the maximum observed plasma concentration (tmax)
time of last quantifiable concentration | 72 hours
  time of last quantifiable concentration (Tlast)
• percentage of extrapolated AUC0-∞ | 72 hours
  percentage of extrapolated AUC0-∞ (%AUCextrap)
terminal elimination half-life | 72 hours
  terminal elimination half-life(T1/2)
apparent clearance | 72 hours
  apparent clearance (CL/F)
apparent volume of distribution | 72 hours
  apparent volume of distribution (VZ/F)
amount excreted in urine | 72 hours
  amount excreted in urine (Ae)
percentage excreted in urine | 72 hours
  percentage excreted in urine (Fe)
renal clearance | 72 hours
  renal clearance (CLR)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - At Fort Lauderdale Behavioral Health Center, Oakland Park, Florida
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com